CLINICAL TRIAL: NCT06502431
Title: Analysis of Disturbances in Neurofluid Dynamics in Type I Chiari Malformations
Acronym: NEUROFLUX-C
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PI2023_843_0033
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Type I Chiari Malformation; Cerebral Hemodynamic; Craniospinal Hydrodynamic; Phase Contrast MRI; Cerebrospinal Fluid
Keywords: Type I Chiari Malformation; Cerebral hemodynamic; Craniospinal hydrodynamic; Phase contrast MRI; Cerebrospinal fluid
MeSH Terms: conditions — Arnold-Chiari Malformation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Symptomatic CMI group (Experimental)
  Interventions: Other: phase contrast sequences
- Non-Symptomatic CMI group (Experimental)
  Interventions: Other: phase contrast sequences
- Control group (Active Comparator)
  Interventions: Other: phase contrast sequences

INTERVENTIONS:
Other: phase contrast sequences — patients will benefit from phase contrast sequences complementary to the morphological MRI performed as part of the patient management.

SUMMARY:
A global analysis of craniospinal hemodynamics and hydrodynamics is necessary to better understand the pathophysiology of Chiari malformations. This includes an analysis of intraventricular CSF flow, intracranial subarachnoid spaces, foramen magnum, cervical subarachnoid spaces and within the syringomyelia cavity when present. The investigators will also analyze the pulsatility of the cerebellar tonsils in the foramen magnum. Hemodynamic analysis will be performed at the high cervical level (internal carotid and vertebral arteries, jugular veins) and intracranially (carotid and basilar arteries, right sinus and superior longitudinal sinus). This analysis will be made possible by PCMRI acquisitions with slice planes allowing the analysis of the dynamics of the CSF (mesencephalic aqueduct, prepontic cisterns, foramen magnum, at the level of the C2C3 disc, syringomyelia if present), cerebellar tonsils (foramen magnum). The cross-sectional planes for hemodynamic analysis will be at the level of the C2C3 disc (cervical vascular analysis) and upstream of the polygon of Willis (intracranial vascular analysis).

The goal is to complement the clinical and morphological investigations with quantitative imaging of cerebrospinal fluid (CSF) and blood flow in the craniospinal system. These flows are potentially altered or causes of this Chiari anomaly.

The investigators propose a translational research project of clinical research allowing the analysis of a diagnostic technique by a diagnostic, monocentric, prospective study. After neurosurgical consultation, patients with Chiari malformation will be assigned to a symptomatic Chiari malformation or a non-symptomatic Chiari malformation group. They will be offered to participate in this study after information and informed consent. The allocation between the two groups will be made according to the symptomatic or non-symptomatic nature of the Chiari malformation. After inclusion, the patients will have a morphological MRI and a PCMRI according to the determined slice plans and allowing a global analysis of the craniospinal hemohydrodynamics. Craniospinal hemohydrodynamics in a control population will also be analyzed using the same methodology by PCMRI.

ELIGIBILITY:
Inclusion Criteria:

* All patients with major symptomatic or nonsymptomatic CMI
* aged 18 to 50 years
* no previous neurosurgical, neurological, or cardiological history.
* Controls should be age-matched to symptomatic CMI group. They should not have a history of neurosurgery, neurology, or cardiology.

Exclusion Criteria:

* Patients who are minors or over 50 years of age
* CMI invalidated by our radiological review
* Neurosurgical, neurological or cardiological history
* MRI contraindication
* pregnant, breast-feeding and parturient women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
CSF Flow | day 1
  Flow will be measured by the oscillatory volume expressed in mL/cardiac cycle.
Blood Flow | day 1
  Flow will be measured by the oscillatory volume expressed in mL/cardiac cycle.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No